CLINICAL TRIAL: NCT04627857
Title: Effect of the Use of Specific Oral Hygiene Devices on Gingival Health Among Patients With Systemic Sclerosis
Acronym: ScleroBross
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8014
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Scleroderma Systemic
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Manual toothbrush (Active Comparator)
  Interventions: Device: Manual toothbrush
- Arm 2: Manual toothbrush and water flosser (Philips Sonicare AirFloss Ultra) (Experimental)
  Interventions: Device: Manual toothbrush and water flosser (Philips Sonicare AirFloss)
- Arm 3: Manual toothbrush and water flosser (Philips Sonicare AirFloss Ultra) (Experimental)
  Interventions: Device: Sonic toothbrush
- Arm 4: Sonic toothbrush (Philips Sonicare ProtectiveClean) and water flosser (Experimental)
  Interventions: Device: Sonic toothbrush (Philips Sonicare) and water flosser (Philips Sonicare AirFloss)

INTERVENTIONS:
Device: Manual toothbrush — Patients in group 1 (''reference procedure'') receive a manual toothbrush with a small compact head to facilitate access to the posterior teeth and soft bristles.
  Arms: Arm 1: Manual toothbrush
Device: Manual toothbrush and water flosser (Philips Sonicare AirFloss) — - Group 2 patients receive a manual toothbrush with a small, compact head for easy access to the posterior teeth and soft bristles. They also receive a Philips brand interdental microjet (Philips Sonicare AirFloss Ultra) which must be filled with water.
  Arms: Arm 2: Manual toothbrush and water flosser (Philips Sonicare AirFloss Ultra)
Device: Sonic toothbrush — - Group 3 patients receive a rechargeable sonic electric toothbrush from Philipps with an integrated excess pressure sensor and a compact toothbrush head for easy access to the posterior teeth.
  Arms: Arm 3: Manual toothbrush and water flosser (Philips Sonicare AirFloss Ultra)
Device: Sonic toothbrush (Philips Sonicare) and water flosser (Philips Sonicare AirFloss) — - Group 4 patients receive a Philips Sonicare ProtectiveClean rechargeable sonic electric toothbrush with an integrated excess pressure sensor and 2 compact toothbrush heads for easy access to the posterior teeth. They also receive an interdental microjet from Philips (Philips Sonicare AirFloss Ultra) which must be filled with water.
  Arms: Arm 4: Sonic toothbrush (Philips Sonicare ProtectiveClean) and water flosser

SUMMARY:
Systemic sclerosis is a rare multisystem connective-tissue disorder characterized by three major pathological hallmarks: widespread fibrosis, vasculopathy and immunological abnormalities. This condition has multiple effects on the orofacial region that is involved in approximately 80% of the patients with a significant impact on the quality of life.

The aim of this randomized single-blind study is to evaluate the impact of the use of a specific oral hygiene instrumentation (sonic toothbrush and water flosser with a large handle) compared to "standard" toothbrushing with a manual toothbrush on the gingival health among patients with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female ≥ 18 years (18th birthday completed)
* Affiliation to a social welfare system
* Signed informed consent form
* More than 12 natural teeth suitable for evaluation
* Systemic sclerosis with cutaneous involvement with a diagnosis based on American College of Rheumatology (ACR) and LeRoy and Metzger criteria

Exclusion Criteria:

* Localized scleroderma or systemic sclerosis without cutaneous involvement ("sine scleroderma" limited form)
* Less than 12 natural teeth suitable for evaluation and/or mandibular/maxillary complete denture(s)
* Other progressive chronic illness /autoimmune disease other than systemic sclerosis (e.g. diabetes)
* Another cause of mucocutaneous sclerosis (e.g. radiotherapy involving the oro-facial region)
* Current use of sonic toothbrush and/or dental water flosser
* Severe manual handicap preventing the patient from holding a toothbrush with a large handle
* Oral antiseptics (e.g. chlorhexidin mouthwashes)
* Ongoing medical treatment inducing a significant modification of the gingival state (e.g. anti-epileptic drugs)
* Smoking (≥ 10 cigarettes per day)
* Impossibility to provide accurate information (e.g. emergency situation, comprehension difficulties)
* Individual under guardianship, curatorship or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Changing of plaque index between baseline, week 2 and week 4 | day 0, week 2 and week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Service de parodontologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No